CLINICAL TRIAL: NCT00664547
Title: Reduction in Cardiovascular Risk Factors and Visceral Adipose Tissue in Men: Separate Effects of Diet- and Exercise-Induced Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Queen's University
Model: Parallel | Purpose: Treatment
Other Study IDs: Ross 1997
Record Dates: First submitted 2008-04-21; First posted 2008-04-23 (Estimated); Last update posted 2008-04-23 (Estimated); Status verified 2008-04

CONDITIONS: Obesity
Keywords: obesity, exercise, diet, insulin resistance
MeSH Terms: conditions — Obesity; Motor Activity; Insulin Resistance | interventions — Diet, Reducing; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- C (No Intervention)
- DWL (Active Comparator): Diet Weight Loss
  Interventions: Behavioral: Diet Weight Loss
- EWL (Active Comparator): Exercise Weight Loss
  Interventions: Behavioral: Exercise Weight Loss
- EWS (Active Comparator): Exercise without weight loss
  Interventions: Behavioral: Exercise Without Weight Loss

INTERVENTIONS:
Behavioral: Diet Weight Loss
  Arms: DWL
Behavioral: Exercise Weight Loss
  Arms: EWL
Behavioral: Exercise Without Weight Loss
  Arms: EWS

SUMMARY:
The purpose of the trial was to examine the independent effects of equivalent diet- or exercise-induced weight loss on obesity and related cardiovascular health risk factors. We hypothesized that exercise would result in greater reductions in obesity and health risk factors that equivalent diet (caloric restriction).

ELIGIBILITY:
Inclusion Criteria:

* Men between 20 and 60 yrs

Exclusion Criteria:

* Smokers and diabetics

Ages: 20 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 1997-09; Primary Completion 1999-12 (Actual); Study Completion 1999-12 (Actual)

PRIMARY OUTCOMES:
Abdominal obesity | 3 months
Insulin Resistance | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert Ross, PhD, Principal Investigator — Queen's University
Locations (1):
- Queen's University, Kingston, Ontario, Canada

REFERENCES:
- [Result] Ross R, Dagnone D, Jones PJ, Smith H, Paddags A, Hudson R, Janssen I. Reduction in obesity and related comorbid conditions after diet-induced weight loss or exercise-induced weight loss in men. A randomized, controlled trial. Ann Intern Med. 2000 Jul 18;133(2):92-103. doi: 10.7326/0003-4819-133-2-200007180-00008. PMID 10896648